CLINICAL TRIAL: NCT06483269
Title: Homologus PRP in the Infiltrative Treatment of Knee Osteoarthritis in Young Athletic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP-Sport Pilot
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infiltrative procedure (Other)
  Interventions: Procedure: PRP infiltration

INTERVENTIONS:
Procedure: PRP infiltration — a single intra-articular infiltration of 5 mL of PRP-O will be performed by the infiltrating physician.
  It is specified that the PRP-O used within the study will be produced following the guidelines and standards for the production of blood products for non-transfusion use as already in place at the Unified Metropolitan Transfusion Service IOR site.
  PRP (Platelet Rich Plasma) is produced from platelet pool from donor buffy coat.
  PRP contains 1,000,000 PLT/mml +/- 20%, as required by current regulations.

SUMMARY:
The study consists of 3 phases (enrollment, infiltrative procedure, and controls):

* Identification by specialized orthopedic medical staff belonging to the SC Orthopedic and Trauma Clinic II of the Rizzoli Orthopedic Institute of subjects who meet the study inclusion criteria. Signing of informed consent form and completion of evaluation questionnaires.
* infiltrative procedure
* Patients will be clinically evaluated before the infiltration procedure and at 1, 3, 6, and 12 months after treatment by trained medical personnel (outcome assessors). Questionnaires will be administered for clinical evaluations before treatment and at these clinical checkups during follow-up. Any adverse events to treatment will also be assessed during follow-up visits. The duration and extent of joint swelling and pain following infiltration will be reported, and any drug therapies taken by the patient will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients, both sexes, with symptomatic knee osteoarthritis with:
* Age: 18-40 years;
* Unilateral involvement;
* Signs and symptoms of knee osteoarthritis;
* Radiographic or MRI signs of degenerative pathology of knee cartilage (Kellgren-Lawrence grade 1-3);
* Ability and consent of patients to actively participate in clinical follow-up;
* Signature of informed consent;
* Pain ≥ 4 on VAS s

Exclusion Criteria:

* Patients unable to express consent;
* Patients undergoing intra-articular infiltration of other substance in the previous 6 months;
* Patients undergoing knee surgery in the previous 12 months;
* Patients with malignant neoplasms;
* Patients with rheumatic diseases;
* Patients with uncontrolled metabolic diseases;
* Patients with hematological diseases (coagulopathies);
* Patients abusing alcoholic beverages, drugs or medications;
* Knee trauma treated in the previous 6 months.
* Other conditions that may interfere with the evaluation of OA treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee score | 6 months
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function.

SECONDARY OUTCOMES:
International Knee Documentation Committee score | baseline, 1, 3, 6, 12 months
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function.
Tegner Activity Level Scale | baseline, 1, 3, 6, 12 months
  It is a questionnaire to find out the patient's level of physical activity
Knee Injury and Osteoarthritis Outcome Score | baseline, 1, 3, 6, 12 months
  The full questionnaire consists of five subscales and they cover: pain (9 items), symptoms (7 items of which two relate to stiffness), functions and activities of daily living (17 items) physical function, sports activities and leisure (5 items) and quality of life in relation to the knee (4 items). All items in the relevant subscales have the same response mode, use a 5-point Likert scale, and each question is assigned a score from 0 to 4, where 0 indicates "no difficulty" and 4 "a severe difficulty). Score range 0-100 for each subscale.
Visual Analogue Scale | baseline, 1, 3, 6, 12 months
  visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable"
objective parameter | baseline, 1, 3, 6, 12 months
  range of motion and bilateral trans patellar and supra patellar circumferences for comparative analysis.
Patient Acceptable Symptom State | baseline, 1, 3, 6, 12 months
  Valuable tool for assessing patient satisfaction considering the patient's current degree of pain, function, and daily activity.
Expectations of treatment efficacy | baseline
  The patient should indicate at baseline what benefits he or she expects from the treatment.
Overall judgment on treatment | baseline, 1, 3, 6, 12 months
  The patient should indicate the degree of satisfaction related to the treatment performed at each follow-up.

OTHER OUTCOMES:
Tolerability assessment parameters: | baseline, 1, 3, 6, 12 months
  All adverse events will be reported by filling out "Adverse event report forms" that will be kept with each patient's CRF (Case Report Form). The latter will document all medications taken additionally by the patient for pain control, indicating brand name, generic name, start and end of intake, and daily dose.
  Serious adverse events will be reported as per company procedure and the Ethics Committee will be informed, which will rule on whether patient enrollment should be discontinued.
Platelet-rich plasma-Homologous (PRP-O) evaluation parameters | baseline, 1, 3, 6, 12 months
  The quality of the administered Platelet-rich plasma- Homologous (PRP-O) will be assested by using standard blood parameters data as hematological control.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS - Istituto ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Everts PA, Knape JT, Weibrich G, Schonberger JP, Hoffmann J, Overdevest EP, Box HA, van Zundert A. Platelet-rich plasma and platelet gel: a review. J Extra Corpor Technol. 2006 Jun;38(2):174-87. PMID 16921694
- [Result] Sanchez AR, Sheridan PJ, Kupp LI. Is platelet-rich plasma the perfect enhancement factor? A current review. Int J Oral Maxillofac Implants. 2003 Jan-Feb;18(1):93-103. PMID 12608674